CLINICAL TRIAL: NCT02801422
Title: Altered Neural Activation Patterns of Emotional Processing in Dependent Cannabis Users Associated With Relapse
Brief Title: Neural Indices Associated With Relapse in Cannabis Dependence
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University of Electronic Science and Technology of China (Other)
Collaborators: German Research Foundation (Other); University Hospital, Bonn (Other)
Responsible Party: Principal Investigator, Benjamin Becker, Prof. Dr. rer. nat. Benjamin Becker, University of Electronic Science and Technology of China
Other Study IDs: ART_Can_03
Record Dates: First submitted 2016-06-11; First posted 2016-06-15 (Estimated); Last update posted 2018-10-29 (Actual); Status verified 2018-10

CONDITIONS: Cannabis Dependence
Keywords: cannabis; fMRI; addiction; relapse
MeSH Terms: conditions — Marijuana Abuse; Behavior, Addictive; Recurrence

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Cannabis Dependence: ages 18-40
  Interventions: Other: fMRI
- Healthy control subjects: socio-demographically matched
  Interventions: Other: fMRI

INTERVENTIONS:
Other: fMRI

SUMMARY:
The aim of this fMRI study is to investigate neural indices of relapse in cannabis dependence. The development and maintenance of drug addictions have been associated with deficits in cognitive control, craving and impaired stress regulation. Therefore, neural markers of brain processes underlying the beforementioned components will be studied. Subsequent follow-up drug use interviews will reveal associations between relapse in cannabis dependence and alterations in brain networks of cognitive control, craving and stress.

ELIGIBILITY:
Inclusion Criteria:

* Cannabis Dependence
* 24 hours abstinence

Exclusion Criteria:

* other DSM-4 diagnosis
* neurological disorder

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Cannabis dependent individuals
Sampling Method: Non-Probability Sample
Enrollment: 75 (Estimated)
Dates: Start 2016-02; Primary Completion 2019-03 (Estimated); Study Completion 2019-03 (Estimated)

PRIMARY OUTCOMES:
fMRI neural activation patterns of emotional processing | one time point = fMRI assessment after minimum 24 hours of abstinence
  Activation patterns associated with emotion processing, emotion regulation, craving and stress are determined in addicted cannabis users compared to non-using matched control subjects

SECONDARY OUTCOMES:
Timeline Followback Interviews | one time point = 12 months after fMRI data acquisition
  Association between fMRI correlates and drug use during follow up preiod as predictor for relapse

CONTACTS AND LOCATIONS:
Locations (1):
- University of Bonn, Bonn, North Rhine Westfalia, Germany